CLINICAL TRIAL: NCT00366600
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HKI-272 Administered Orally to Healthy Subjects.
Brief Title: Study Evaluating HKI-272 Administered to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-107
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Breast Cancer; Health; Pharmacokinetics; healthy subjects
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib

INTERVENTIONS:
Drug: neratinib — HKI-272

SUMMARY:
Safety and tolerability of HKI-272 in healthy subjects; the influence of food intake on the same.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2006-07; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics; safety and tolerability; influence of food on the same.

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- Northwest Kinetics, Tacoma, Washington, United States